CLINICAL TRIAL: NCT03182881
Title: Effectiveness of Myofascial Release Versus Manual Lymphatic Drainage After Breast Cancer Surgery In Women Undergoing Conservative Surgery and Radiotherapy. Randomized Clinical Trial
Brief Title: Effectiveness of Myofascial Release Versus Manual Lymphatic Drainage After Breast Cancer Surgery
Acronym: MRvsMLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Dr, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0016
Record Dates: First submitted 2017-06-03; First posted 2017-06-09 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Fibromyalgia
Keywords: Myofascial-reléase; Fibromyalgia; Lymphatic drainage; Breast cancer
MeSH Terms: conditions — Fibromyalgia; Breast Neoplasms | interventions — Manual Lymphatic Drainage; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miofascial-reléase (Experimental): Myofascial Release (MR), with the purpose of releasing fascial restriction zones and major fibrosis (thoraco-brachial) caused by restriction after CM tto. IM therapy was applied to the affected area. The position of the patient was identical during both treatment sessions.
  Interventions: Other: Myofascial Release
- Manual Lymphatic Drainage (MLD) (Active Comparator): It was applied following the Leduc method with the patient in a supine position with 30º elevation of the arm and very superficial and smooth maneuvers were performed in the axillary lymph nodes, in the chest region and in the arm with the same sequence as Guerero et al. The objective of the application in our study is to obtain a beneficial treatment for the patient since it produces an increase of blood and lymphatic circulation, with positive effects on the peripheral vegetative nervous system.
  Interventions: Other: Lymphatic Drainage

INTERVENTIONS:
Other: Lymphatic Drainage — It was applied with the patient in a supine position with 30º elevation of the arm and very superficial and smooth maneuvers were performed in the axillary lymph nodes, the chest region and the arm.
  Arms: Manual Lymphatic Drainage (MLD)
Other: Myofascial Release — For the use of the treatment the bases of Pilat, A. 2016 were followed. The global and specific techniques for the periganglionar and upper thoracic region were chosen. The application of each smooth maneuver three-dimensional fascial movement has been carried out has an approximate duration of about 10 minutes and a total of 50 minutes.
  Arms: Miofascial-reléase

SUMMARY:
Objective. To compare the effectiveness of myofascial therapy against manual lymphatic drainage in the reduction of sequelae secondary to conservative surgery and radiotherapy in women who survived breast cancer.

Design. Randomized clinical trial. Site. Faculty of Physiotherapy of the University of Valencia. Participants. Twenty-four patients were included in the study. Interventions. 13 patients were randomly assigned to treatment with myofascial therapy and 11 to receive manual lymphatic drainage.

Main measurements. Pain measured using the Visual Analogue Scale, shoulder joint range, shoulder functionality using the DASH questionnaire, quality of life assessed using the FACT-B questionnaire, and the depressed status of the patients using the PHQ-9 . All of this was assessed before and after treatment, and one month later as follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30 and 60 diagnosed with breast cancer undergoing conservative / partial surgery.
* Without lymphedema or mild lymphedema.
* They must have finished the coadjuvant treatment.

Exclusion Criteria:

* Women with muscle or tendon lesions in the arm.
* Kin disorders or circulatory pathology.
* Chemotherapy or radiotherapy.
* Surgical history in the area are excluded from the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Pain | 2 months
  The Visual Analog Scale (EVA) was used. This scale consists of marking on a horizontal line of 10 cm in length VAS is a 10-point rating scale (0 = absolute discomfort and 10 = full comfort).

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy Breast | 2 months
  Consists of 36 items separated into two components: a general one formed by the first 27 items, and a specific one related to the symptoms of breast cancer constituted by the remaining 9 items. The survey represents five domains: physical well-being (7 items), social and family welfare (7 items), emotional well-being (6 items), functional well-being (7 items) and a specific subscale related to breast cancer and its treatment.
Disabilities of the Arm, Shoulder and Hand (DASH) | 2 months
  The Functional Assessment of Cancer Therapy Breast (FACT-B). This questionnaire is a specific instrument for assessing quality of life related to upper limb problems. It consists of 30 items, which assess situations of daily life and the patient responds by giving a score to each item that ranges from 1 "no difficulty", 2 "Little difficulty", 3 "Moderate difficulty", 4 "Very difficult" and 5 "Unable".
Joint mobility | 2 months
  The measurement of the angular travel of all the movements of the shoulder was evaluated through a universal goniometer which proved to be a valid and reliable instrument.
Depressive state | 2 months
  Evaluated using the patient's health questionnaire-9 (PHQ-9). It consists of 9 items that assess the presence of depressive symptoms during the last two weeks. The score range is 0-27, each item ranges from 0 (never) to 3 (more than half the days).

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma Victoria Espí López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serra-Ano P, Ingles M, Bou-Catala C, Iraola-Lliso A, Espi-Lopez GV. Effectiveness of myofascial release after breast cancer surgery in women undergoing conservative surgery and radiotherapy: a randomized controlled trial. Support Care Cancer. 2019 Jul;27(7):2633-2641. doi: 10.1007/s00520-018-4544-z. Epub 2018 Nov 24. PMID 30470892